CLINICAL TRIAL: NCT03231124
Title: A Phase 1, Single Centre Randomised, Double-blind Placebo-controlled Multiple Dose Study With Incremental Dosing to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral Doses of LEO 32731 in Healthy Male Japanese Subjects.
Brief Title: Multiple Dose Study With Incremental Dosing to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral Doses of LEO 32731 in Healthy Male Japanese Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0058-1362; 2017-000907-26 (EudraCT Number)
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: LEO 32731 and Placebo tablets are of identical appearance. The packaging and labelling of the IMPs and Placebo contain no evidence of their identity. It is not considered possible to differentiate between the IMPs solely by sensory evaluation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LEO 32731 (Experimental): Incremental dosing of LEO 32731 progressing to a maximum of 30 mg.
  * Days 1 - 3: 10 mg dose twice a day for three days
  * Days 4 - 6: 20 mg dose twice a day for three days
  * Days 7 - 11: 30 mg dose twice a day for five days
  * Days 12: 30 mg dose once in the morning
  Interventions: Drug: LEO 32731
- Placebo (Placebo Comparator): Incremental dosing of placebo progressing to a maximum of 30 mg.
  * Days 1 - 3: 10 mg dose twice a day for three days
  * Days 4 - 6: 20 mg dose twice a day for three days
  * Days 7 - 11: 30 mg dose twice a day for five days
  * Days 12: 30 mg dose once in the morning
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LEO 32731 — LEO 32731 is being developed by LEO Pharma.
  Arms: LEO 32731
Drug: Placebo — Placebo contains the same excipients in the same concentration, only lacking LEO 32731
  Arms: Placebo

SUMMARY:
This trial will investigate the safety, tolerability and pharmacokinetic (PK) data of LEO 32731 (and major human metabolite LEO 40815) in healthy male Japanese subjects. The primary objective is the assessment of PK in Japanese subjects.

Data obtained from this trial will be used to compare with existing data from the other Phase 1 trials. This comparison of safety and PK profiles between Japanese and Caucasian subjects will allow the inclusion of Japanese patients into Phase 2b studies.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written, personally signed, and dated informed consent to participate in the study, in accordance with the ICH Good Clinical Practice (GCP) Guideline E6 (1996) and applicable regulations, before completing any study-related procedures.
2. An understanding, willingness and ability to fully comply with study procedures and restrictions.
3. Japanese men aged >20 to <45 years (from date of signing informed consent which is defined as the beginning of the Screening Period). This inclusion criterion will only be assessed at the Screening Visit.
4. Japanese subjects must have lived outside of Japan for ≤ 5 years in total and be first generation Japanese, defined as born in Japan and having 4 biologic grandparents who are ethnic Japanese.
5. Subjects must have a body mass index (BMI) between 18.0-25.0 kg/m².

Exclusion Criteria:

1. Current or recurrent disease (i.e. with, or with a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological, dermatological or other major disorders as determined by the Investigator) that could affect the action, absorption, or disposition of LEO 32731, or could affect clinical assessments or clinical laboratory evaluations.
2. Current or relevant history of physical or psychiatric illness that may require treatment or make the subject unlikely to fully comply with the requirements of the study or complete the study, or any condition that presents undue risk from the investigational product or study procedures.
3. Any history of psychiatric or mental health issue such (including depression) deemed clinically significant as assessed by the Investigator.
4. Any history of/or active cancer or malignancy (other than squamous cell carcinoma more than 5 years prior).
5. History of Wiskott-Aldrich Syndrome
6. History of active tuberculosis, and/or history of partially or incomplete treatment of tuberculosis.
7. Any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, may influence the result of the study, or the subject's ability to participate in the study.
8. Use of any prescribed systemic or topical medication(s) within 14 days or 10 half-lives (whichever is longer) prior to Day 1 of the dosing period.
9. Use of any systemic or topical non-prescribed or over-the-counter (OTC) medication(s) (including multivitamin, herbal, or homeopathic preparations) within 7 days or 5 half-lives (whichever is longer) prior to Day 1 of the dosing period. The occasional use of paracetamol (acetaminophen) is allowed to treat short term adverse events; subject to review by the investigator. The maximum allowed daily dose is 2000 mg for paracetamol at the discretion of the investigator.
10. Consumption of more than 21 units of alcohol per week.
11. History or clinical evidence of substance and/or alcohol abuse within the 12 months before screening. Alcohol abuse is defined as regular weekly intake of more than 21 units for males.
12. Positive test results for alcohol, drugs of abuse at screening or Day -1.
13. Use of tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch) within 90 days prior to Day 1 of the dosing period.
14. Use of an investigational product within 90 days prior to Day 1 of the dosing period or active enrolment in another drug or vaccine clinical study.
15. Known or suspected intolerance, hypersensitivity or allergy (excluding non-active hayfever) to any drug, food or other known substance (including investigational product, its closely related compounds, and/or any of the stated ingredients).

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from zero to 12 hour (AUC0-12) on day 12 of LEO 32731. | on Day 12
Time to reach maximum observed plasma concentration (tmax) on day 12 of LEO 32731. | on Day 12
Maximum observed plasma concentration (Cmax) on day 12 of LEO 32731. | on Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Lorch, MD, Principal Investigator — Richmond Pharmacology
Locations (1):
- Investigational Site, London, United Kingdom